CLINICAL TRIAL: NCT04930484
Title: Cultural Adaptation, Validity and Reliability of the Turkish Version of Performance Measure for Activities of Daily Living-8
Brief Title: Validity and Reliability of the Turkish Version of Performance Measure for Activities of Daily Living-8
Status: Completed | Type: Observational
Sponsor: Ahi Evren Chest and Cardiovascular Surgery Education and Research Hospital (Other)
Responsible Party: Principal Investigator, NUREL ERTURK, Doctora student, Ahi Evren Chest and Cardiovascular Surgery Education and Research Hospital
Other Study IDs: GO 20/1171
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Congestive Heart Failure
Keywords: Congestive heart failure; Functional limitation; Questionnaire
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic heart failure (CHF) is characterized by limited exercise performance, which is mainly determined by disease-specific factors, such as diminished cardiac output, abnormal ventilatory response, and low perfusion in skeletal muscles, which lead to skeletal muscle dysfunction.1 Exercise intolerance and symptoms may lead to activity restriction and further functional deterioration with the progression of CHF. There is some evidence that disease-specific self-report measures more quantify clinically relevant domains than measures of general health status and are generally more sensitive to clinical change. aim of the study is to investigate the validity and reliability of the PMADL-8 questionnaire in the Turkish population.

DETAILED DESCRIPTION:
Chronic heart failure (CHF) is characterized by limited exercise performance, which is mainly determined by disease-specifi factors, such as diminished cardiac output, abnormal ventilatory response, and low perfusion in skeletal muscles, which lead to skeletal muscle dysfunction.Exercise intolerance and symptoms may lead to activity restriction and further functional deterioration with the progression of CHF.

There is some evidence that disease-specific self-report measures more quantify clinically relevant domains than measures of general health status and are generally more sensitive to clinical change. aim of the study is to investigate the validity and reliability of the PMADL-8 questionnaire in the Turkish population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 45-75 years, who are conscious, able to answer all questions, can communicate in Turkish, diagnosed with CHF, have NYHA (New York Heart Association) heart failure functional classification II and III and agree to participate in the study will be included in the study.

Exclusion Criteria:

* CHF patients with NYHA functional class IV who were hospitalized, who are unable to cooperate, and not willing to participate.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample size of the study was determined as at least 40 people, 5 times the number of items used in the scale.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Performance Measure For Activities Of Daily Living-8 | 6 month
  The questionnaire consists of 8 questions. It is a daily living activities measurement questionnaire consisting of 4 categories (very easy = 1 point, easy = 2, difficult = 3 points, very difficult = 4 points). High scores indicate severe functional limitations.
Chronic Heart Failure Questionnaire | 6 month
  The questionnaire consists of 20 questions and four sub-dimensions. The sub-dimensions of the scale are dyspnea (5 questions), fatigue (4 questions), mood (7 questions) and dominance (4 questions). The questions have Likert-type response options ranging from 1 (worst) to 7 (best). The higher the score, the higher the quality of life.
Nothingham Health Profile | 6 month
  It is a general health questionnaire consisting of 6 sub-parameters consisting of energy level (ES), emotional reactions (ER), physical activity (FA), pain (A), sleep (U) and social isolation (SI) and a total of 38 items.
Sociodemographic data form | 6 month
  Gender, age, height, weight, body mass index, complaints, concomitant diseases, smoking and alcohol history, New York Heart Association's (NYHA) Congestive Heart Failure Classification, Coronary Artery Disease Risk Factors (Kwong et al. Circulation 2003) will be questioned. . Shortness of breath (at rest and on exertion) will be assessed with the modified Borg Scale

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Nurel, Akçaabat, Trabzon
  - Trabzon Ahi Evren Thoracic and Cardiovascular Surgery Training and Research Hospital, Trabzon

IPD SHARING:
Plan to Share IPD: No